CLINICAL TRIAL: NCT04714944
Title: Gut Microbial Substrate Switch to Improve Metabolic Health
Brief Title: Fiber and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL72483.068.20
Record Dates: First submitted 2020-12-04; First posted 2021-01-20 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): isocaloric placebo
  Interventions: Dietary Supplement: Placebo
- whole fiber product (Experimental): 15 g for 2 weeks, followed by 30 g for 10 weeks
  Interventions: Dietary Supplement: Whole fiber product

INTERVENTIONS:
Dietary Supplement: Placebo — Supplementation period 12 weeks
  Arms: Placebo
Dietary Supplement: Whole fiber product — Supplementation period 12 weeks
  Arms: whole fiber product

SUMMARY:
Based on previous research of the investigators group, the investigators hypothesize that slowly fermentable fibers with a high degree of polymerization that increase SCFA specifically in the distal colon are expected to have higher potential for influencing host metabolism and metabolic health by improving adipose tissue function, preventing lipid overflow and hepatic as well as skeletal muscle fat accumulation thereby improving insulin sensitivity.

The objective of this randomized clinical trial is to test, whether the a dietary fiber product containing different physiological acting fibers reverses peripheral and hepatic insulin resistance in overweight/obese insulin resistant participants.

ELIGIBILITY:
Inclusion criteria:

Overweight/obese insulin resistant/prediabetic participants (age 45-70 y, BMI ≥ 28 kg/m2 < 35 kg/m2)

Exclusion criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L and 2h glucose ≥ 11.1 mmol/L)
* Gastroenterological diseases or abdominal surgery;
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than 5 years;
* Abuse of products; alcohol and drugs, excessive nicotine use defined as >20 cigarettes per day;
* Plans to lose weight or following of a hypocaloric diet;
* Regular supplementation of pre- or probiotic products, use of pre- or probiotics 3 months prior to the start of the study;
* Intensive exercise training more than three hours a week;
* Use of any medication that influences glucose or fat metabolism and inflammation (i.e. NSAIDs);
* Regular use of laxation products;
* Use of antibiotics in the last three months (antibiotics use can alter substantially the gut microbiota composition).
* Follow a vegetarian diet.
* Metal objects such as implants present in the body (e.g. electronic implants, pacemakers, metal fragments in the eyes, skin or body)
* The use of permanent make-up (eyeliners, eyebrows) or tattoos on the head, shoulders, breast or neck
* Claustrophobia

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | Before and 12 week after the start of the intervention
  The change of peripheral insulin sensitivity as assessed by a hyperinsulinaemic-euglycemic clamp

SECONDARY OUTCOMES:
hepatic and adipose tissue insulin sensitivity | Before and 12 week after the start of the intervention
  The change in hepatic and adipose tissue insulin sensitivity as assessed by a hyperinsulinaemic-euglycemic clamp
Energy expenditure (indirect calorimetry) | Before and 12 week after the start of the intervention
  The change in energy expenditure as measured via ventilated hood system
Substrate oxidation (indirect calorimetry) | Before and 12 week after the start of the intervention
  The change in substrate oxidation as measured via ventilated hood system
Faecal and circulating SCFA | Before and 12 week after the start of the intervention
  The change in faecal and circulating SCFA
Faecal microbiota composition and in vitro microbial activity testing | Before and 12 week after the start of the intervention
  The change in faecal microbiota composition as assessed via 16s rRNA gene sequencing
In vitro microbial activity testing | Before and 12 week after the start of the intervention
  The change in fin vitro microbial activity testing as assessed using an in vitro model of the human colon
Circulating hormones such as insulin | Before and 12 week after the start of the intervention
  The change in circulating hormones in peripheral blood
Circulating metabolites such as glucose | Before and 12 week after the start of the intervention
  The change in metabolites in peripheral blood
Circulating inflammatory markers such as TNF | Before and 12 week after the start of the intervention
  The change in inflammatory markers in peripheral blood
body weight | Before and 12 week after the start of the intervention
  The change in body weight in kg
body composition | Before and 12 week after the start of the intervention
  The change in body compostion as assessed using DEXA scans
liver fat content | Before and 12 week after the start of the intervention
  The change in liver fat content as assessed by proton magnetic resonance spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Omary L, Canfora EE, Puhlmann ML, Gavriilidou A, Rijnaarts I, Holst JJ, Op den Kamp-Bruls YMH, de Vos WM, Blaak EE. Intrinsic chicory root fibers modulate colonic microbial butyrate-producing pathways and improve insulin sensitivity in individuals with obesity. Cell Rep Med. 2025 Jul 15;6(7):102237. doi: 10.1016/j.xcrm.2025.102237. PMID 40669445